CLINICAL TRIAL: NCT05719285
Title: Single-Dose Versus Multi-Dose Prophylactic Antibiotic Administration for Bladder OnabotulinumtoxinA Injection
Brief Title: Prophylactic Antibiotic Administration for Bladder OnabotulinumtoxinA Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-698
Record Dates: First submitted 2023-01-23; First posted 2023-02-08 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-09

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome; Urge Incontinence; Urinary Incontinence, Urge
Keywords: incontinence; overactive bladder; urge incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Anti-Bacterial Agents; Antibiotic Prophylaxis

STUDY DESIGN:
Intervention Model Description: Men and women 18 years of age or older with refractory overactive bladder or neurogenic bladder will be randomized in a 1:1 ratio into one of two groups until the targeted sample size is met:
  * The single dose group will receive one dose of antibiotic prior to intradetrusor Botox injection.
  * Individuals in the multi-dose group will receive one dose of antibiotic prior to intradetrusor Botox injection and additional antibiotics for a total of three days of antibiotic administration.
  Random permuted block randomization with block sizes of 2, 4, 6, and 8 will be used to assign eligible patients to treatment groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1: Single-Dose Antibiotic Prophylaxis (Active Comparator): Patients will receive one dose of antibiotic prior to bladder onabotulinumtoxinA injection.
  Interventions: Drug: Single-Dose Antibiotic
- 2: Multi-Dose Antibiotic Prophylaxis (Active Comparator): Patients will receive one dose of antibiotic prior to bladder onabotulinumtoxinA injection. The same antibiotic will be continued for 3 days of total antibiotic administration with additional doses prescribed to the patient's pharmacy.
  Interventions: Drug: Multi-Dose Antibiotic

INTERVENTIONS:
Drug: Single-Dose Antibiotic — Allergy, prior urine culture resistance or another contraindication to first line antibiotic will result in the patient being prescribed second line antibiotic and so forth.
  First line:
  Arm 1: trimethoprim / sulfamethoxazole 800/160 mg once pre-procedure
  Second line:
  Arm 1: cefalexin 500 mg once pre-procedure
  Third line:
  Arm 1: nitrofurantoin 100 mg once pre-procedure
  Fourth line:
  Arm 1: ciprofloxacin 500 mg once pre-procedure
  Other Names: ARM 1: Single-Dose Antibiotic Prophylaxis
  Arms: 1: Single-Dose Antibiotic Prophylaxis
Drug: Multi-Dose Antibiotic — Allergy, prior urine culture resistance or another contraindication to first line antibiotic will result in the patient being prescribed second line antibiotic and so forth.
  First line:
  Arm 2: trimethoprim / sulfamethoxazole 800/160 mg once pre-procedure plus 800/160 mg every twelve hours for 6 total doses
  Second line:
  Arm 2: cefalexin 500 mg once pre-procedure plus 500 mg every twelve hours for 6 total doses
  Third line:
  Arm 2: nitrofurantoin 100 mg once pre-procedure plus 100 mg every twelve hours for 6 total doses
  Fourth line:
  Arm 2: ciprofloxacin 500 mg once pre-procedure plus 500 mg every twelve hours for 6 total doses
  Other Names: ARM 2: Multi-Dose Antibiotic Prophylaxis
  Arms: 2: Multi-Dose Antibiotic Prophylaxis

SUMMARY:
The goal of this clinical trial is to evaluate the outcomes of differing durations of antibiotic prophylaxis with bladder onabotulinumtoxinA injection in patients with refractory overactive bladder.

The main question it aims to answer are:

• Is the incidence of post-procedure UTI similar between single-dose and multi-day durations of peri-procedural antibiotics?

Participants will be randomized to single-dose versus multi-day dose of antibiotic prophylaxis with bladder onabotulinumtoxinA injection.

Researchers will compare incidence of UTI in each group to see if there is a significant difference.

DETAILED DESCRIPTION:
* After informed consent is obtained, urinalysis will be collected. Post-void residual will also be assessed by bladder scan if not already documented in the electronic medical record in the prior three months.
* Patients with positive urinalysis and symptomatic for UTI will be excluded from the study.
* Patients will be randomized in a 1:1 ratio to one of two groups.

  * Group 1 will receive one dose of antibiotic prior to bladder onabotulinumtoxinA injection.
  * Group 2 will receive one dose of antibiotic prior to bladder onabotulinumtoxinA injection.
  * The same antibiotic will be continued for 3 days of total antibiotic administration with additional doses prescribed to the patient's pharmacy.
* Bladder onabotulinumtoxinA injection and dosing will be completed based on the surgeon's standard technique and template.
* Bladder onabotulinumtoxinA injection will be completed by staff or fellows in the Female Pelvic Medicine and Reconstructive Surgery division of the Genitourinary and Kidney Institute.
* Patients will be followed for 4 weeks after the procedure.
* At 4 weeks study investigators will contact the patient by phone to evaluate for any UTIs or adverse events not previously reported by the patient during the study period.
* Chart review will occur at 4 weeks to assess for any unreported events.
* Other than this additional phone call, post-operative patient management will not deviate from the standard of care.
* Patients will be instructed to report symptomatic UTIs, urinary retention, or any other adverse events related to onabotulinumtoxinA or antibiotic to investigators.
* Patients that report symptoms suggestive of a UTI will result in obtaining a urine culture.
* Symptomatic, culture proven UTIs will be treated with appropriate antibiotics per the current AUA guidelines.
* Symptoms suggestive of urinary retention, such as increased urinary frequency, voiding small amounts of urine, or feelings of incomplete bladder emptying, will result in obtaining a post void residual (PVR) and urinalysis.
* Patients will undergo teaching to perform self, clean intermittent catheterization of the bladder per the discretion of the operating surgeon.
* Any adverse reactions to the prescribed antibiotic will result in discontinuation of the antibiotic and managed according to the severity of the reaction.

Antibiotic regimens:

Allergy, prior urine culture resistance or another contraindication to first line antibiotic will result in the patient being prescribed second line antibiotic and so forth.

First line:

Group 1: trimethoprim / sulfamethoxazole 800/160 mg once pre-procedure Group 2: trimethoprim / sulfamethoxazole 800/160 mg once pre-procedure plus 800/160 mg every twelve hours for 6 total doses

Second line:

Group 1: cefalexin 500 mg once pre-procedure Group 2: cefalexin 500 mg once pre-procedure plus 500 mg every twelve hours for 6 total doses

Third line:

Group 1: nitrofurantoin 100 mg once pre-procedure Group 2: nitrofurantoin 100 mg once pre-procedure plus 100 mg every twelve hours for 6 total doses

Fourth line:

Group 1: ciprofloxacin 500 mg once pre-procedure Group 2: ciprofloxacin 500 mg once pre-procedure plus 500 mg every twelve hours for 6 total doses

ELIGIBILITY:
Inclusion Criteria:

* Participants with planned in-office bladder onabotulinumtoxinA injection
* Men or Women Age ≥ 18
* Able to read, speak, and write in English
* No contraindication to injection of onabotulinumtoxinA - hypersensitivity to any botulinum toxin preparation or to any of the components in the formulation
* Willingness and ability to initiate intermittent catheterization post-treatment if required
* No contraindication to oral antibiotics
* No active antibiotic therapy for any indication at the time of onabotulinumtoxinA injection
* Have not participated in this study before

Exclusion Criteria:

* Any type of catheterization to empty the bladder
* Unwillingness or inability to initiate intermittent catheterization post-treatment if required
* Less than 3 months since last bladder onabotulinumtoxinA injection
* Pregnant and/or breastfeeding
* Active symptomatic UTI the day of the procedure - new or worsening frequency, urgency, dysuria, hematuria, suprapubic/flank pain, fevers or chills
* History of recurrent UTI
* Prior development of urinary retention or incomplete bladder emptying after bladder onabotulinumtoxinA injection requiring catheterization of any type

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Slopnick, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 1: Single-Dose Antibiotic Prophylaxis: Patients will receive one dose of antibiotic prior to bladder onabotulinumtoxinA injection.
  Single-Dose Antibiotic: Allergy, prior urine culture resistance or another contraindication to first line antibiotic will result in the patient being prescribed second line antibiotic and so forth.
  First line:
  Arm 1: trimethoprim / sulfamethoxazole 800/160 mg once pre-procedure
  Second line:
  Arm 1: cefalexin 500 mg once pre-procedure
  Third line:
  Arm 1: nitrofurantoin 100 mg once pre-procedure
  Fourth line:
  Arm 1: ciprofloxacin 500 mg once pre-procedure
- 2: Multi-Dose Antibiotic Prophylaxis: Patients will receive one dose of antibiotic prior to bladder onabotulinumtoxinA injection. The same antibiotic will be continued for 3 days of total antibiotic administration with additional doses prescribed to the patient's pharmacy.
  Multi-Dose Antibiotic: Allergy, prior urine culture resistance or another contraindication to first line antibiotic will result in the patient being prescribed second line antibiotic and so forth.
  First line:
  Arm 2: trimethoprim / sulfamethoxazole 800/160 mg once pre-procedure plus 800/160 mg every twelve hours for 6 total doses
  Second line:
  Arm 2: cefalexin 500 mg once pre-procedure plus 500 mg every twelve hours for 6 total doses
  Third line:
  Arm 2: nitrofurantoin 100 mg once pre-procedure plus 100 mg every twelve hours for 6 total doses
  Fourth line:
  Arm 2: ciprofloxacin 500 mg once pre-procedure plus 500 mg every twelve hours for 6 total doses
Period: Overall Study
Arm/Group | 1: Single-Dose Antibiotic Prophylaxis | 2: Multi-Dose Antibiotic Prophylaxis
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Single-Dose Antibiotic Prophylaxis | 2: Multi-Dose Antibiotic Prophylaxis | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Full Range); unit: years] | 69.42 [28 to 87] | 64.62 [30 to 93] | 67.02 [30 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 50 | 96
  Male | 4 | 0 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 32.26 [18.56 to 70.53] | 34.14 [19.73 to 75.86] | 33.20 [18.56 to 75.86]
Current Anti-Cholinergic Use [Number; unit: participants] | 7 | 7 | 14
Prior Anti-Cholinergic Use [Number; unit: participants] | 41 | 41 | 82
Current Beta-3 Agonist Use [Number; unit: participants] | 6 | 7 | 13
Prior Beta-3 Agonist Use [Number; unit: participants] | 24 | 22 | 46
Current Posterior Tibial Nerve Stimulation (PTNS) Use [Number; unit: participants] | 0 | 0 | 0
Prior Posterior Tibial Nerve Stimulation (PTNS) Use [Number; unit: participants] | 3 | 1 | 4
Current Sacral Neuromodulation Use [Number; unit: participants] | 4 | 4 | 8
Prior Sacral Neuromodulation Use [Number; unit: participants] | 4 | 5 | 9
Previous Bladder Botox [Number; unit: participants] | 39 | 38 | 77
Neurogenic Bladder [Number; unit: participants] | 2 | 1 | 3
Current Vaginal Estrogen use [Number; unit: participants] — Population: Vaginal estrogen status is only assessed in female patients
  participants
    number analyzed (Participants) | 46 | 50 | 96
    (all) | 4 | 8 | 12
Diabetes Mellitus [Count of Participants; unit: Participants] | 14 | 13 | 27
Current Tobacco Use [Number; unit: participants] | 6 | 4 | 10
Sleep Apnea [Number; unit: participants] | 22 | 10 | 32

OUTCOME MEASURES:

1. Primary Outcome: Establish Noninferiority of the Single Dose Antibiotic Administration to the Multi-dose Antibiotic Administration.
Description: To assess this aim, the rate of postoperative urinary tract infection (UTI) within 4 weeks following bladder onabotulinumtoxinA injection will be compared between groups. Noninferiority will be declared if the incidence of UTI in the single dose group is not more than UTI incidence in the multiple dose group within statistical variability, by the prespecified noninferiority margin.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1: Single-Dose Antibiotic Prophylaxis | 2: Multi-Dose Antibiotic Prophylaxis
Number analyzed (Participants) | 50 | 50
Participants | 1 | 1

2. Secondary Outcome: Antibiotic Adverse Events
Description: Summarize rates of adverse events related to antibiotics in each group.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1: Single-Dose Antibiotic Prophylaxis | 2: Multi-Dose Antibiotic Prophylaxis
Number analyzed (Participants) | 50 | 5
Participants | 0 | 0

3. Secondary Outcome: Symptomatic Urinary Retention
Description: Estimate the rate of symptomatic urinary retention requiring catheterization among refractory overactive bladder patients who experience a UTI.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1: Single-Dose Antibiotic Prophylaxis | 2: Multi-Dose Antibiotic Prophylaxis
Number analyzed (Participants) | 50 | 50
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Patients will be instructed to report symptomatic UTIs, urinary retention, or any other adverse events related to onabotulinumtoxinA or antibiotic to investigators. At 4 weeks study investigators will contact the patient by phone to evaluate for any UTIs or adverse events not previously reported by the patient during the study period. Chart review will occur in 4 weeks to assess any unreported events.
Arm/Group | 1: Single-Dose Antibiotic Prophylaxis | 2: Multi-Dose Antibiotic Prophylaxis
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/50
Other Adverse Events (participants affected / at risk) | 4/50 | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Single-Dose Antibiotic Prophylaxis (N=50) | 2: Multi-Dose Antibiotic Prophylaxis (N=50)
Cellulitis (Infections and infestations) | 0 | 1 (1) — A disorder characterized by an infectious process involving the skin such as cellulitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1: Single-Dose Antibiotic Prophylaxis (N=50) | 2: Multi-Dose Antibiotic Prophylaxis (N=50)
Bronchial Infection (Infections and infestations) | 1 (1) | 0 (0) — A disorder characterized by an infectious process involving the bronchi
Cystitis noninfective (Renal and urinary disorders) | 2 (2) | 1 (1) — Microscopic hematuria; minimal increase in frequency, urgency, dysuria, or nocturia; new onset of incontinence
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) — A disorder characterized by laboratory test results that indicate blood in the urine.
Urinary Retention (Renal and urinary disorders) | 2 (2) | 1 (1) — A disorder characterized by accumulation of urine within the bladder because of the inability to urinate.
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 2 (2) — A disorder characterized by an infectious process involving the urinary tract, most commonly the bladder and the urethra.
Urinary Tract Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) — A disorder characterized by blockage of the normal flow of contents of the urinary tract
Vaginal Infection (Infections and infestations) | 0/46 (0) | 1 (1) — A disorder characterized by an infectious process involving the vagina.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT05719285/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT05719285/ICF_001.pdf